CLINICAL TRIAL: NCT02629783
Title: Psychomotor Therapy as Complimentary Treatment to Patients With Shoulder Pain - a Randomized Controlled Trial.
Brief Title: Psychomotor Therapy as Complimentary Treatment to Patients With Shoulder Pain.
Acronym: PsychShoP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-20150111
Record Dates: First submitted 2015-11-24; First posted 2015-12-14 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Physical Therapy Modalities; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy + Corticosteroid injection + Psychomotor therapy (Experimental): Usual care + intervention
  Interventions: Other: Psychomotor therapy; Other: Physiotherapy; Drug: corticosteroid injection
- Physiotherapy + Corticosteroid injection (Active Comparator): Usual care
  Interventions: Other: Physiotherapy; Drug: corticosteroid injection

INTERVENTIONS:
Other: Psychomotor therapy — 1 treatment of approximately 45 minutes the first 5 weeks after randomization. The treatment will focus on teaching the patients about body awareness and handling of there shoulder problems in daily living.
  Arms: Physiotherapy + Corticosteroid injection + Psychomotor therapy
Other: Physiotherapy — Patients are, in secondary care setting, given 3-5 basic physiotherapy exercises for there shoulder pain, targeting rotator cuff muscles and scapula thoracic muscles. Furthermore they are given advice on seeking further physiotherapy guidance in private setting.
Drug: corticosteroid injection — At baseline, patients with signs of inflammation in the subacromial bursa, can receive a ultrasound guided corticosteroid injection in the bursa

SUMMARY:
Some patients with shoulder pain have decreased body awareness (BA). To some degree, pain among these patients can be increased due to their lack in BA. Psychomotor therapy is thought to improve BA and thereby increase the effect of traditional therapy, such as physiotherapy and exercises.

The aim of this study is therefore to investigate if psychomotor therapy, as a complimenting treatment to physiotherapy, decreases shoulder patients' function deficits and pain reported on PRO's, compared to physiotherapy alone.

DETAILED DESCRIPTION:
Study design:

This trial, is a randomised, controlled, observer-blinded superiority trial, with a two-group parallel design, to be conducted in Denmark. The primary endpoint will be 12 weeks after baseline. Patients will be randomised to either "Intervention+Usual Care" or "Usual Care" (block randomization with a 1:1 allocation).

Settings and locations:

Patients will be recruited from the shoulder unit at the outpatient clinic, orthopaedic department at Hospital Lillebaelt - Vejle Hospital.

Randomisation and allocation concealment:

Patients will be randomly assigned to either of the two groups with a 1:1 allocation as per a computergenerated randomisation schedule, stratified by administration of concomitant corticosteroid injection using permuted blocks of random sizes (two to six). The primary investigator, assessors and administrator of the randomisation procedure will not know block sizes in order to ensure allocation concealment

Blinding:

Outcome assessors will perform both baseline and followup assessments, and will be kept blinded from treatment allocation. At the follow-up assessments, patients will be strongly encouraged not to disclose the components of their intervention programme, in order to keep the outcome assessor blinded.

Statistical analysis plan:

The primary efficacy analysis performed is assessment of the between-group difference in change in the DASH score after 12 weeks in the intent-to-treat (ITT) population (all randomised patients independent of compliance and withdrawals). In the case of missing data due to dropouts, a non-responder imputation will be applied; a baseline observation carried forward (BOCF) technique will be used for patients who do not complete the study. For the primary analyses at week 12, we will use analysis of covariance (ANCOVA) to compare the progressive high-load exercise group with the low-load exercise group for mean changes from baseline in the DASH score, as well as the secondary continuous outcomes. The primary model includes the change from baseline as the dependent variable, with treatment group (Intervention OR Usual care), corticosteroid status (yes or no) as main effects, with the baseline score as an additional covariate.

To analyse the longitudinal element of time effects of NRS in the randomized trial (repeated measures design 1-24 weeks), a linear approach will be used, fitted in SAS software (version 9.3 Service Pack 4; SAS Institute Inc., Cary, North Carolina, United States) using the procedure 'PROC MIXED' based on restricted maximum likelihood (REML) estimates of the parameters. The variable 'patient' will be applied as a random effects factor. Assessment of the treatment and time effects is of exploratory interest for the primary outcome in testing for a possible interaction, and both treatment and time will be used as systematic factors, using the baseline value as covariate to reduce random variation and increase power.

ELIGIBILITY:
Inclusion Criteria:

* >three months of should pain
* Disturbed sleep due to shoulder pain
* VAS resting pain above 2 OR VAS activity pain above 5
* MAIA score <= 3
* Read and understand Danish.

Exclusion Criteria:

* Frozen shoulder
* Glenohumeral (GH) arthritis
* Rotator Cuff (RC) rupture
* GH instability
* Acromioclavicular joint arthritis
* Operation in the shoulder joint within the last six months
* Cervical problems
* Psychiatric diagnosis
* Alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Patient reported function and pain on the "Disability in the Arm, Shoulder and Hand (DASH) questionnaire" | Change from baseline DASH at 12 weeks
  Patient reported generic shoulder outcome questionnaire (questions upon function and pain related limitations).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression score (HAD) | Change from baseline HAD at 12 weeks
  Patient reported generic mental outcome measure
Hospital Anxiety and Depression score (HAD) | Change from baseline HAD at 24 weeks
  Patient reported generic mental outcome measure
Pain on the NRS Scale | Change from baseline NRS at weeks 1-24
  "Short Message Service" (SMS) is sent to the patients phone regarding pain.
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Change from baseline MAIA at 12 weeks
  Patient reported generic body awareness outcome measure
Multidimensional Assessment of Interoceptive Awareness (MAIA) | Change from baseline MAIA at 24 weeks
  Patient reported generic body awareness outcome measure

OTHER OUTCOMES:
Quality of life on "EQ-5D" | Change from baseline EQ-5D at 12 weeks
  Patient reported generic quality of life outcome measure
Quality of life on "EQ-5D" | Change from baseline EQ-5D at 24 weeks
  Patient reported generic quality of life outcome measure
Patient reported function and pain on the "Disability in the Arm, Shoulder and Hand (DASH) questionnaire" | Change from baseline DASH at 24 weeks
  Patient reported generic shoulder outcome questionnaire (questions upon function and pain related limitations).

CONTACTS AND LOCATIONS:
Overall Officials: Lilli Soerensen, MD, Study Chair — Outpatient shoulder clinic, orthopaedic department at Hospital Lillebaelt - Vejle Hospital; Kim G. Ingwersen, PhD.Fellow, Principal Investigator — Rehabilitation department at Hospital Lillebaelt - Vejle Hospital
Locations (1):
- Shoulder clinic, Orthopedic department, Hospital Lillebaelt - Vejle Hospital, Vejle, Jutland, Denmark

REFERENCES:
- [Derived] Ingwersen KG, Vobbe JW, Pedersen LL, Sorensen L, Wedderkopp N. Effect of Psychomotricity in Combination With 3 Months of Active Shoulder Exercises in Individuals With Chronic Shoulder Pain: Primary Results From an Investigator-Blinded, Randomized, Controlled Trial. Arch Phys Med Rehabil. 2019 Nov;100(11):2136-2143. doi: 10.1016/j.apmr.2019.05.032. Epub 2019 Jun 24. PMID 31247165